CLINICAL TRIAL: NCT04872751
Title: The Malaysian Study On Hemodialysis Patients SARS-COV-2 Vaccination Immune Response: A Prospective Observational Cohort Study
Brief Title: Immune Response of Haemodialysis Patients Post Covid-19 Vaccination
Acronym: Covid-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Penang Hospital, Malaysia (Other Government)
Responsible Party: Principal Investigator, Dr.Ong Loke Meng, Doctor, Penang Hospital, Malaysia
Other Study IDs: NMRR-21-634-59445
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Immune Response Post Covid 19 Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess immune response of end stage renal failure patients after Covid 19 vaccination

ELIGIBILITY:
Inclusion Criteria:

* ESRF patient on hemodialysis who are eligible for the goverment Covid 19 vaccination programme
* 18 years old and above
* consented to join the study

Exclusion Criteria:

* patient who refused to be vaccinated
* patient who deemed unsuitable for Covid vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage renal failure (ESRF) receiving hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 425 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in post vaccination SARS-CoV-2 neutralizing antibody level | up to one year
  Study the antibody synthesis induced by vaccination, among end stage renal failure patients, and the change in its level at 1 month, at 6 months and at 1 year after complete vaccination.

SECONDARY OUTCOMES:
Change From Baseline in post vaccination SARS-CoV-2 neutralizing antibody level after 1st inoculation of the vaccine (incomplete vaccination) | one month
  Study the antibody synthesis and the change in its level after 1st inoculation of the vaccine

CONTACTS AND LOCATIONS:
Overall Officials: LokeMeng Ong, Principal Investigator — Penang Hospital
Locations (1):
- Penang Hospital, George Town, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No